CLINICAL TRIAL: NCT05942755
Title: Study of Changes in CSF Ionic Composition After Aneurysmal Meningeal Hemorrhage
Acronym: ION_SAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0245
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid haemorrhage; cerebrospinal fluid; ionic disorders; hyponatremia; normal pressure hydrocephalus; blood-brain barrier; ionogram
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hyponatremia; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subarachnoid haemorrhage with Fisher 3 or 4.: HAS Group :
  * Adults
  * Hospitalized in the neurological intensive care unit for a Fisher 3 or 4 aneurysmal meningeal hemorrhage with external ventricular drain (EVD) and urinary catheter. This EVD allows the evacuation of 10-20ml/h of CSF into an external collector. CSF is usually removed daily.
  * With a catheter (arterial or venous) for repeated sampling. Blood samples are taken as part of routine care on arrival of patients and then every 24 hours if an arterial catheter is in place; otherwise, every Monday, Wednesday and Friday. Samples from the EVD will be taken on Day 0 and then every 24 hours. A urine ionogram is also performed every 24 hours as part of the usual management to regulate water, sodium and potassium intake by enteral or parenteral route.
  In addition, clinical data will be collected every 24 hours on the basis of a computerized medical record without additional examination.
  Interventions: Other: Concurrent evaluation of blood and CSF ionograms to determine if there is a correlation between CSF change and the development of hyoponatremia between day 0 and day 14.
- Control group, normal pressure hydrocephalus: Control group :
  * Adults
  * Performing a perfusion test in the operating room in the context of normal pressure hydrocephalus.
  A lumbar puncture is performed in the operating room to evacuate the chronic CSF effusion in the ventricles (hydrocephalus), before performing an intrathecal perfusion test. 1ml of the CSF thus collected will be analyzed to determine the ionic composition and thus compare it to the CSF collected from patients with SAH.
  Interventions: Other: Concurrent evaluation of blood and CSF ionograms to determine if there is a correlation between CSF change and the development of hyoponatremia between day 0 and day 14.

INTERVENTIONS:
Other: Concurrent evaluation of blood and CSF ionograms to determine if there is a correlation between CSF change and the development of hyoponatremia between day 0 and day 14. — Blood samples are taken as part of routine care on arrival of patients and then every 24 hours if an arterial catheter is in place; otherwise, every Monday, Wednesday and Friday. Samples from the EVD will be taken on Day 0 and then every 24 hours. A urine ionogram is also performed every 24 hours as part of the usual management to regulate water, sodium and potassium intake by enteral or parenteral routine.
  The ionic composition of CSF from patients with SAH will be compared with a control population of patients hospitalized with normal pressure hydrocephalus. A lumbar puncture is performed in the operating room to evacuate the chronic CSF effusion in the ventricles (hydrocephalus), before performing an intrathecal perfusion test. 1ml of the CSF thus collected will be analyzed to determine its ionic composition

SUMMARY:
Hyponatremia is a frequent complication of subarachnoid hemorrhage (SAH) with a prevalence of 30 to 50% in patients with this condition. This hydro-electrolytic disorder is responsible for an increase in morbidity with the appearance of neurological disorders.

Also, it has been shown that there are ionic changes in the cerebrospinal fluid and a probable alteration of the blood-brain barrier in patients with SAH. The kinetics and relationship between hyponatremia and these changes remain unknown.

The main objective of the study is to determine whether the change in cerebrospinal fluid (CSF) composition, precedes the development of hyponatremia. For this, the investigators propose to study the evolution of the CSF ionogram with the blood ionogram. Furthermore, they will perform additional analyses on the basis of a control group (CSF of patient with normal pressure hydrocephalus) to determine the effect of SAH on ionic changes.

The hypothesis of the study is that there is a correlation between the change in CSF blood ionogram and the development of hyponatremia between day 0 and day 14.

ELIGIBILITY:
Inclusion Criteria:

SAH group :

* Adults
* Hospitalized in the neurological intensive care unit for a Fisher modified aneurysmal SAH 3 or 4 with EVD and urinary catheter.
* With a catheter (arterial or venous) for repeated sampling.

Control group :

* Adults
* Performing a perfusion test in the operating room for normal pressure hydrocephalus

Exclusion Criteria:

* Patients with SAH without EVD.
* Patients with non-aneurysmal SAH.
* Pregnant or breastfeeding women.
* Patients under legal protection, guardianship, curatorship, safeguard of justice.
* Patients participating in a study that may interfere with the present study.
* Persons under forced psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SAH group : patients hospitalized in the neurological intensive care with Fisher modified aneurysmal SAH 3 or 4 requiring external ventricular drain.
  Control group : patients hospitalized for normal pressure hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the change in CSF ionogram between day 0 and day 14 according to the occurrence of hyponatremia. | The patient is included during hospitalization within 2 days of the placement of the EVD

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France